CLINICAL TRIAL: NCT07238647
Title: A Phase I, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of Subcutaneous Administration of Single Ascending Doses of HRS-5817 in Obese Participants
Brief Title: A Trial of HRS-5817 in Obese Participants
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5817-103
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: HRS-5817 subcutaneous administration
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: HRS-5817 dose level 1 (Experimental): Single dose of HRS-5817/placebo given subcutaneously (dose level 1)
  Interventions: Drug: HRS-5817
- Experimental: HRS-5817 dose level 2 (Experimental): Single dose of HRS-5817/placebo given subcutaneously (dose level 2)
  Interventions: Drug: HRS-5817
- HRS-5817 dose level 3 (Experimental): Single dose of HRS-5817/placebo given subcutaneously (dose level 3)
  Interventions: Drug: HRS-5817
- HRS-5817 (Experimental): Single dose of HRS-5817/placebo given subcutaneously (dose level 4)
  Interventions: Drug: HRS-5817

INTERVENTIONS:
Drug: HRS-5817 — Single dose of HRS-5817/placebo given subcutaneously (dose level 1 )
  Arms: Experimental: HRS-5817 dose level 1
Drug: HRS-5817 — Single dose of HRS-5817/placebo given subcutaneously (dose level 2 )
  Arms: Experimental: HRS-5817 dose level 2
Drug: HRS-5817 — Single dose of HRS-5817/placebo given subcutaneously (dose level 3 )
  Arms: HRS-5817 dose level 3
Drug: HRS-5817 — Single dose of HRS-5817/placebo given subcutaneously (dose level 4)
  Arms: HRS-5817

SUMMARY:
The purpose of this study is to assess safety, PK, Pharmacodynamic and immunogenicity profile of a single dose of HRS-5817 in obese participants

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 18 to 55 years of age (inclusive)
2. Participants with body mass index (BMI) between 30.0 kg/m2 (inclusive) to 40.0 kg/m2 (inclusive) at screening.
3. Ability to understand the trial procedures and possible adverse events, volunteer to participate in the trial, and provide written informed consent, be able to comply with all the requirements, and able to complete the study.

Negative pregnancy test for women of childbearing potential (WOCBP) at baseline. Men and WOCBP must agree to take highly effective contraceptive methods

Exclusion Criteria:

1. History or evidence of clinically significant disorders 2. Individuals with a weight change of more than 5kg within 3 months prior to the screening.

1. Participant with a history of or current endocrine disorders that may significantly influence body weight (e.g., Cushing's syndrome, hypothyroidism, hyperthyroidism), or with obesity resulting from pharmacotherapy, monogenic mutations, or hereditary obesity syndromes.
2. Any other circumstances (e.g., not suitable for venous access) or laboratory abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.
3. Use of any GLP-1 receptor agonists (including but not limited to Liraglutide, Beneglitide, Semaglutide, and Tirzepatide, etc.) or any other prescription medications, OTC drugs and dietary supplements for weight loss (including but not limited to Orlistat, Naltrexone/Bupropion, Phentermine/Topiramate, ect.). within 3 months prior to screening, and no planned use for the study duration.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Based on Incidence and Severity of Treatment Emergent Adverse Events | Day 253
  Number of participants with Adverse events and Serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Day 253
  Maximum observed plasma concentration (Cmax)
Pharmacokinetics - AUC₀-t | Day 253
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC₀-inf)
Pharmacokinetics - Tmax | Day 253
  Time to reach maximum observed plasma concentration (Tmax)
Pharmacokinetics - t½ | Day 253
  Terminal elimination half-life (t½)
Immunogenicity - Anti-Drug Antibody (ADA) | Day 253
  Incidence and onset time of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Linear, Perth, Western Australia, Australia